CLINICAL TRIAL: NCT05271474
Title: Managing Diagnosed COPD Patients Through Connected Devices to Provide Pulmonologists With Objective Data to Inform Treatment Decisions and Enable Exacerbation Intervention
Brief Title: COPD Remote Patient Monitoring Through Connected Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Innovation Hub Enterprises (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003325
Record Dates: First submitted 2022-02-08; First posted 2022-03-09 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Participants will be assigned to use Sibel sensor and download the ANNE ONE platform to their mobile devices. The Sibel sensors are to be worn on the sternum and index finger and can be attached using provided replaceable gel adhesive. The Sibel sensors will transmit data to the ANNE ONE platform. The ANNE ONE platform will send automated alerts to the CRC via email when a patient is flagged as uncontrolled, which will occur when a patient's vitals reach or pass one of the safety thresholds.
  Interventions: Device: ANNE ONE Platform
- Control Arm (No Intervention): These patients will be followed by the Clinical Research Coordinator for CAT scores, emergency department visits and hospitalizations.

INTERVENTIONS:
Device: ANNE ONE Platform — ANNE ONE is one most advanced digital platforms that are gradually becoming more available to enable providers to help patients manage their condition. It integrates soft and flexible sensors for comprehensive vital signs monitoring. This platform creates objective transparency by automatically recording data from the sensor on the patient, lessening the need for patients to consciously track their COPD exacerbation events, enabling providers to proactively manage their patients' condition, and creating actionable reports for providers to review with their patients.
  Arms: Intervention Arm

SUMMARY:
This study is a device study that will use a double-arm. It will integrate the ANNE ONE platform which continuously tracks enrolled COPD patients' vital signs and symptoms over the course of the study and digitally shares that data with providers for clinical interpretation, potential intervention and treatment decision making and will help evaluate the impact on participating patient's COPD Assessment Test (CAT) scores. Subjects will be recruited from Emory clinics and identified via a data pull based on clinical relevant codes. Letters will be sent out to eligible candidates and interested participants will contact the research team. The research team will consent them over the phone and mail the device to them; participants will be compensated.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a diseases that causes airflow limitation and breathing-related problems, affecting approximately 16 million people in the U.S., most of which are aged 40 and above with a history of smoking. COPD causes acute exacerbations where a patient has worsening symptoms (increased shortness of breath, cough, or sputum production). Managing COPD presents many challenges, as patients struggle to adhere to their prescribed treatment plans. Digital platforms are gradually becoming more available to enable providers to help patients manage their condition. These platforms create objective transparency, lessening the need for patients to consciously track their COPD exacerbation events, enabling providers to proactively manage their patients' condition, and creating actionable reports for providers to review with their patients. Ultimately, connected devices present a strong opportunity to provide patients with appropriate care earlier in the patient journey, while enabling pulmonologists to deliver more customized management based on close to real time objective data.

The primary goal of this study is to evaluate the impact of the implementation of the ANNE ONE platform on patients with COPD's condition. This will be achieved by using the ANNE ONE platform to continuously track enrolled COPD patients' vital signs over the course of the study and digitally sharing that data with providers for clinical interpretation, potential intervention and treatment decision making. Interviews have been conducted with leading pulmonologists and staff at Emory Healthcare to understand what factors are considered when recommending a treatment pathway for a COPD patient, what the current workflow shortcomings are and how a new workflow using the ANNE ONE platform could effectively be integrated at a pulmonologist's office.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40>years
* Have a formal diagnosis of COPD
* Must be able to understand and speak English in order to complete the survey questionnaires.
* They must be able and willing to download the ANNE ONE application on a smartphone.
* Have their COPD managed by a pulmonologist.
* Have the willingness and ability to commit to the study period and completion of the surveys.

Exclusion Criteria:

* Participants with a formal diagnosis of asthma will be excluded.
* Those who are unable to read and/or speak English
* Patients who exhibit physical or mental disability precluding the ability to provide informed consent will be excluded from the study.
* Those who are unable or unwilling to download the ANNE ONE application will also be excluded.
* Additionally, participant who are not willing or able to commit to the duration of the study will not be included.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Exacerbation of COPD episodes by Assessment Test (CAT) scores Changes | At baseline and at 16 weeks
  CRC will be responsible for collecting through patient-reported and electronic medical record (EMR)-reported (clinical notes and/or hospitalizations). Greater impact on COPD Assessment Test (CAT) scores (reduction of patient symptoms) compared to control group.

SECONDARY OUTCOMES:
Number of exacerbations onset detected | From baseline to study completion (16 weeks)
  Clinical Research Coordinators (CRC) will be responsible for collecting through patient-reported and electronical medical record reported (clinical notes and/or hospitalizations).Episodes will be counted and compared from Intervention Group vs Control group.
Vital data: SpO2 drop >4% | From baseline to study completion (16 weeks)
  Data from ANNE ONE sensors will be reviewed for SpO2 drops below 7-day rolling average by more than 4% for 2 consecutive days.
Vital data: SpO2 drop <90% | From baseline to study completion (16 weeks)
  Data from ANNE ONE sensors will be reviewed for SpO2 drops below 90% for 2 consecutive days.
Vital data: FEV1 | From baseline to study completion (16 weeks)
  Data from ANNE ONE sensors will be reviewed for Forced expiratory volume in the first second (FEV1) drops below 7-day rolling average by more than 1.645 standard deviations for 2 consecutive days.
Vital data: Respiratory Rate | From baseline to study completion (16 weeks)
  Data from ANNE ONE sensors will be collected reviewed for respiratory rate increases 15% for 2 consecutive days above 7-day rolling average.
Provider Satisfaction Scores | Week 16
  CRC will connect with pulmonologists throughout the pilot and provide a closing survey
Change in Patient Satisfaction Scores | Week 16
  CRC will distribute survey to patients, once at the end of the pilot to understand patient experience and adherence.
Number of Patient Emergency Visits | Week 16
  CRC will be responsible for patient history surveys, as well as coordinating an electronical medical record for the population. CRC will keep up with emergency visits for each subject and record these.
Number of Uncontrolled Flags | From baseline to study completion (16 weeks)
  Number of events that the system shows as "irregular" readings
Response to Flags | From baseline to study completion (16 weeks)
  Number of response received by providers to flags in the system triggered by patient's irregular readings

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Velasquez, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No